CLINICAL TRIAL: NCT00255905
Title: Is Insomnia a Modifiable Risk Factor for Major Depressive Disorder
Brief Title: Cognitive Behavioral Therapy for the Treatment of Depression-Related Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21MH067184 (NIH); R21MH067184 (NIH); DATR A2-AID
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Depression
Keywords: Depression; Insomnia
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) for insomnia
Behavioral: Clinician monitoring

SUMMARY:
This study will determine the effectiveness of cognitive behavioral therapy (CBT) in treating insomnia symptoms that are secondary to depression. This study will also determine how long the benefits of CBT will last and how the recurrence of insomnia is associated with the onset of new depressive episodes.

DETAILED DESCRIPTION:
Insomnia, characterized by an inability to initiate and maintain sleep, is a defining feature of mood disorders such as depression. CBT has been found to be an effective treatment for depression-related insomnia. This study will determine the effectiveness of CBT in treating insomnia that is secondary to depression. In addition, this study will assess the relationship between insomnia and depression, since previous studies have shown that insomnia may not only be a symptom of depression but may also indicate the onset of a depressive episode.

Participants will be randomly assigned to receive weekly sessions of either CBT or clinician monitoring for 8 weeks. Participants in both groups will meet with a therapist at selected visits, but only CBT participants will receive actual therapy. All participants will have 13 study visits; four will be overnight visits in a sleep lab. On Visit 1, participants will complete questionnaires about their sleep quality and symptoms of depression. Participants will also undergo a physical exam and will begin a daily sleep diary. Visits 2, 3, 12, and 13 will be overnight visits in the sleep lab. During these visits, participants will have electrodes placed on their bodies and a polysomnograph will be used to monitor their sleep. Participants will meet with their therapist on Visits 4 to 11. Participants' sleep diaries, depression scales, and sleep scales will be used for assessment. After the intervention part of the study is complete, participants will have monthly follow-up visits for up to 2 years. During the follow-up visits, participants will complete questionnaires about their sleep quality and symptoms of depression.

ELIGIBILITY:
Inclusion Criteria:

* History of recurrent depression with the age of onset between 20 and 40 years of age
* At least one depressive episode within 2 years prior to study entry
* At least three discrete depressive episodes within 10 years prior to study entry
* Successful treatment for or resolution of last episode of depression
* Participants whose depression is in remission are eligible for study enrollment. Criteria for remission includes more than 3 consecutive weeks during which the patient does not meet DSM-IV criteria for depression; a Hamilton Rating Depression Scale score less than 6 and a Beck Depression Inventory (BDI) less than 6; no feelings of depression for at least 6 months prior to study entry; and have not taken depression medication for at least 3 months prior to study entry. Once enrolled in the study, these participants must score less than 6 on the weekly BDIs for the first 3 weeks of the study.
* Have experienced mental stability between depressive episodes
* Willing to discontinue over-the-counter or naturopathic remedies for insomnia or depression during the study
* Able to write and speak English fluently

Exclusion Criteria:

* Current use of maintenance antidepressant therapy
* History of a failure to respond to citalopram treatment
* Unstable medical or psychiatric illness other than major depressive disorder
* History of seizures or head injury
* Current substance or alcohol abuse
* Symptoms suggestive of sleep disorders other than insomnia
* Pregnancy or plan to become pregnant within 2 years of study entry

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2004-07; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Treatment outcome of patients receiving CBT compared to clinician monitoring

SECONDARY OUTCOMES:
Association between rapid eye movement (REM) latency and treatment outcome

CONTACTS AND LOCATIONS:
Overall Officials: Michael Perlis, PhD, Principal Investigator — University of Rochester Sleep Research Lab; Michael Privitera, MD, Principal Investigator — Department of Psychiatry, University of Rochester
Locations (1):
- University of Rochester Sleep and Neurophysiology Research Lab, Rochester, New York, United States

REFERENCES:
- [Background] Perlis ML, Smith MT, Orff H, Enright T, Nowakowski S, Jungquist C, Plotkin K. The effects of modafinil and cognitive behavior therapy on sleep continuity in patients with primary insomnia. Sleep. 2004 Jun 15;27(4):715-25. doi: 10.1093/sleep/27.4.715. PMID 15283007
- [Background] Smith MT, Perlis ML, Park A, Smith MS, Pennington J, Giles DE, Buysse DJ. Comparative meta-analysis of pharmacotherapy and behavior therapy for persistent insomnia. Am J Psychiatry. 2002 Jan;159(1):5-11. doi: 10.1176/appi.ajp.159.1.5. PMID 11772681